CLINICAL TRIAL: NCT06597617
Title: Persistent Organic Pollutants and Mechanical Discharge: Limiting the Impact of Bariatric Surgery Through Personalized Adapted Physical Activity
Acronym: PERSIST-APA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-PP-03
Record Dates: First submitted 2024-07-17; First posted 2024-09-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Control (No Intervention)
- GEA (Aerobic training) (Experimental)
  Interventions: Behavioral: Adapted physical activity with aerobic training [GEA]
- GRM (Strength training) (Experimental)
  Interventions: Behavioral: Adapted physical activity with strength training [GRM]

INTERVENTIONS:
Behavioral: Adapted physical activity with aerobic training [GEA] — Participants will be required to take part in 3 weekly sessions of adapted physical activity for 3 months following bariatric surgery. These sessions (not exceeding 1 hour and 10 minutes) will focus on aerobic training. The first 3 sessions will be accompanied, and will take place either by videoconference or face-to-face, depending on the patient's wishes. Thereafter, each 1st session of the following weeks will also be accompanied and carried out either by videoconference or face-to-face. The following 2 sessions of the week will be carried out autonomously.
  Each session will be organized into (i) a 5-minute cardio-respiratory warm-up and joint mobilization, (ii) a block of aerobic activity and (iii) a 2-minute cool-down including breathing exercises. Training will take place in 2 phases. The first phase will involve a total of 90 minutes of aerobic training spread over 3 sessions. The second phase will involve a total of 150 minutes of aerobic training over 3 sessions.
  Arms: GEA (Aerobic training)
Behavioral: Adapted physical activity with strength training [GRM] — Participants will be required to take part in 3 weekly sessions of adapted physical activity for 3 months following bariatric surgery. These sessions (not exceeding 1 hour and 10 minutes) will focus on eccentric training. The first 3 sessions will be accompanied and conducted face-to-face. Thereafter, each 1st session of the following weeks will also be accompanied and carried out face-to-face. The following 2 sessions of the week will be carried out autonomously.
  Each session will be organized into (i) a 5-minute cardio-respiratory warm-up and joint mobilization, (ii) muscle-strengthening exercises and (iii) a 2-minute cool-down including breathing exercises. The exercises used will mainly involve the lower limbs. Training will take place in 2 phases. The first phase will involve an exposure/adaptation phase to eccentric training. The second phase will involve a gradual increase in intensity.
  Arms: GRM (Strength training)

SUMMARY:
For the most severe cases of obesity, recourse to bariatric surgery is the ultimate solution. Although highly beneficial to individual health, this massive loss of body mass could also have negative effects on metabolism and neuromuscular function. Unfortunately, these effects have been relatively little studied in the scientific literature, and are poorly taken into account in patient follow-up when bariatric surgery has been recommended. One of the adverse effects of bariatric surgery is the release into the bloodstream of Persistent Organic Pollutants (POPs) which, are not only persistent, but also bioaccumulative, toxic and mobile. The major problem is that these circulating POPs are linked to a number of adverse side effects, including reproductive disorders, neurobehavioral alterations, metabolic disorders, gut microbiota alterations inflammatory changes and physiological alterations. POP neurotoxicity could also affect psychomotor abilities and neuromuscular function. In addition, the mechanical unloading (i.e., reduced mechanical stress on muscles) induced by loss of body mass, an effect targeted by bariatric surgery and largely beneficial to the health of individuals, could also alter neuromuscular function and potentially alter muscle architecture and contractile properties. Unfortunately, no data are currently available in the scientific literature to confirm or refute these hypotheses. Physical activity-based intervention strategies may be usefull to counteract the effects of mechanical unloading and the release of POPs as suggested in scientific literature. However it is also possible to question which exercise modality should be preferred. Our hypothesis is that eccentric muscle strengthening would better preserve muscle mass and neuromuscular function while limiting the risks associated with POPs release, compared with an aerobic and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18-55 years)
* Patient scheduled for bariatric surgery
* Patient practicing a leisure-time physical activity < 8 hours of moderate intensity per week or < 4 hours of high intensity per week
* Presence of effective contraception (hormonal or mechanical)

Exclusion Criteria:

* Patient already involved in another experimental study
* Pregnant (urine pregnancy test) or breast-feeding women
* Patient in a particular situation deemed incompatible with the study by the investigator
* Patients from outside the Alpes-Maritimes and Var departments
* Patient having received antibiotic treatment during the 3 months preceding the first stool collection
* Presence of a contraindication to adapted physical activity
* Presence of a contraindication to neurostimulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
MVC (Maximum Voluntary Contraction) | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Unit used to quantify MVC (Maximum Voluntary Contraction): Nm. Description: MVC will be obtained using an ergometer and force sensors.
Blood concentration for each POP investigated | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Unit used to quantify blood concentration for each POP (Persistent Organic Pollutant) investigated: ng/g of lipid.

SECONDARY OUTCOMES:
Total POPs blood concentration [∑POPs] | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Total POPs blood concentration [∑POPs] (ng/ml) will be obtained with the analysis of a blood sampling by chromatography and spectrometry.
Quantity by POPs category | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Quantity by POPs category (ng/ml) will be obtained with the analysis of a blood sampling by chromatography and spectrometry.
Specific and relative muscle strength | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Specific and relative muscle strength (N m) will be obtained using an ergometer and force sensors.
M-wave | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  M-wave will be obtained using an EMG device.
NAV [Voluntary Activation Level] | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  NAV [Voluntary Activation Level] (%) will be obtained using an ergometer, force sensors and a stimulator device
Fatigability | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Fatigability (Δ N m) will be obtained using an ergometer, force sensors and a muscular fatigue protocol.
Pennation angle | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Pennation angle (°) will be obtained by muscle ultrasound imaging.
Muscle thickness | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Muscle thickness (mm) will be obtained by muscle ultrasound imaging.
Fascicle length | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Fascicle length (mm) will be obtained by muscle ultrasound imaging.
Characterization of gut microbiota | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Alpha and beta diversity will be obtained by the analysis of feces collected with specific sampling kit.
Weight | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Weigh (kg) will be obtained by using a weight balance.
Fat mass | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Fat mass (kg and %) will be obtained by using an impedancemeter.
Lean mass | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Lean mass (kg and %) will be obtained by using an impedancemeter.
Body mass index (BMI) | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Body mass index (kg/m^2) will be obtained by using weight balance and a height chart.
Waist-to-hip ratio | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Waist-to-hip ratio will be obtained by measuring the waist circumference (cm) and the hip circumference (cm) with the WHO protocol.
Total cholesterol | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Total cholesterol (g/l) will be obtained with blood sampling analysis.
Free cholesterol | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Free cholesterol (g/l) will be obtained with blood sampling analysis.
Total intra-serum lipids | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Total intra-serum lipids (g/l) will be obtained with blood sampling analysis.
Phospholipids | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Phospholipids (g/l) will be obtained with blood sampling analysis.
Triglycerides | One week prior to bariatric surgery, 1 month after bariatric surgery, 4 months after bariatric surgery and 12 months after bariatric surgery.
  Triglycerides (g/l) will be obtained with blood sampling analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CHEVALIER, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No